CLINICAL TRIAL: NCT04931849
Title: A Pilot Study of Avatrombopag for Temozolomide-induced Thrombocytopenia in Glioma (APATIT-G)
Brief Title: Study of Avatrombopag for Temozolomide-induced Thrombocytopenia in Glioma (APATIT-G)
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI and Sponsor decided to not proceed with the trial.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Frank Akwaa, Assistant Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCS20154
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Thrombocytopenia
Keywords: Thrombocytopenia; Temozolomide; Avatrombopag; Temozolomide-induced Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Avatrombopag (Experimental): Avatrombopag 40 mg daily by mouth (PO)
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — Avatrombopag is a small molecule thrombopoeitic receptor agonist (TPO-RA) that mimics the biological effects of thrombopoeitin (TPO)

SUMMARY:
The purpose of this study is to determine if using avatrombopag in patients with thrombocytopenia due to temozolomide treatment can safely improve a patient's platelet count and allow the patient to complete the temozolomide treatment course as planned.

DETAILED DESCRIPTION:
The purpose of this study is to determine if using avatrombopag in patients with low platelet count due to temozolomide treatment is safe, while at the same time assess whether the avatrombopag can improve the low platelet count and allow the temozolomide treatment to continue as planned.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of grade 2, 3 or 4 glioma
* Subject has initiated concurrent RT and temozolomide followed by planned 6-12 cycles of temozolomide;
* Subject is willing and able to provide written informed consent;
* Subject is ≥ 18 years of age at the time of informed consent;
* Subject is willing and able to comply with all aspects of the protocol;
* Subject had platelet counts ≥ 100, 000/uL at the start of RT+TMZ or TMZ alone;
* Subject experienced grade ≥ 3 (moderate to severe) thrombocytopenia, defined by platelet counts ≤ 50 x 109/L, measured at least 24 hours apart, during the induction RT+TMZ, or at any time during the maintenance TMZ;
* Subject is able to continue to receive temozolomide regimen at the standard maintenance dose and schedule;
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
* Subject has a life expectancy > 12 weeks at screening and is able to receive at least 2 additional cycles of TMZ;
* Females of childbearing potential must agree to use a highly effective method of contraception (combination of condom, diaphragm, or sponge with a spermicide) throughout the entire study period and for 28 days after the investigational product (IP) discontinuation;

Exclusion Criteria:

* History of hematologic malignancy, including leukemia, myeloma, myeloproliferative disease, lymphoma, or myelodysplastic syndrome;
* Subject with history of solid tumor and has received chemotherapy alone or chemotherapy and radiation in the past 5 years;
* Subject has received > 2 previous lines of chemotherapy;
* Subjects who have previously received radiation treatments to the pelvic region including brachytherapy;
* Subject with an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 x upper limit of normal (ULN) or total bilirubin ≥ 3 x upper limit of normal;
* Subject is known to be human immunodeficiency virus positive;
* Known clinically significant acute or active bleeding (e.g., gastrointestinal or central nervous system) within 7 days of screening;
* Known history of thrombophilia with high risk of thrombosis (e.g., homozygous factor V Leiden mutation or prothrombin G20210A mutation, anti-thrombin deficiency, protein C deficiency, protein S deficiency, or antiphospholipid antibody syndrome);
* Subject has a medical condition that, in the opinion of the investigator, would compromise the subject's ability to safely complete the study, such as unstable angina, renal failure requiring dialysis, or active infection requiring intravenous antibiotics;
* History of arterial or venous thrombosis within 6 months of screening;
* Subject has used vitamin K antagonist within 7 days of screening (use of low molecular weight heparin, factor Xa inhibitors, or direct thrombin inhibitors is allowed);
* Subject has a history of chronic platelet or bleeding disorder or thrombocytopenia due to another etiology other than temozolomide (e.g., chronic liver disease or immune thrombocytopenia purpura);
* Subject has used moderate or strong dual inducer of cytochrome P450 (CYP) 2C9 or CYP3A4/5 such as rifampin within 7 days of screening, and/or moderate or strong dual inhibitor such as fluconazole;
* Subject has previously received a thrombopoietin receptor agonist (e.g., eltrombopag or romiplostim) for the treatment of temozolomide induced thrombocytopenia;
* Subject has received a platelet transfusion within 3 days of screening;
* Subject is unable to take oral medication;
* Female subjects who are lactating or pregnant at screening (as documented by positive serum beta-human chorionic gonadotropin [β-hCG] test) or the baseline visit (serum pregnancy test);
* For all men and women of childbearing potential: Refusal or inability to use effective means of contraception;
* History of significant cardiovascular disease or arrhythmia known to increase the risk of thromboembolic events such as atrial fibrillation, coronary artery stent placement, angioplasty, or coronary artery bypass graft) within 6 months of screening;
* Subject is currently enrolled in another clinical study with any investigational drug or device within 30 days of screening; however, participation in observational studies is permitted;
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2024-07-18 (Estimated)

PRIMARY OUTCOMES:
Safety of treatment | 48 weeks
  Measure of time from study enrollment until progression.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided